CLINICAL TRIAL: NCT02452294
Title: An Open-label, Uncontrolled, Single Arm Phase II Trial of Buparlisib in Patients With Metastatic Melanoma With Brain Metastases Not Eligible for Surgery or Radiosurgery
Brief Title: Buparlisib in Melanoma Patients Suffering From Brain Metastases (BUMPER)
Acronym: BUMPER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120ZDE01T
Record Dates: First submitted 2015-05-05; First posted 2015-05-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Malignant Melanoma; Metastases
Keywords: Brain
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buparlisib (Experimental): Patients will receive oral buparlisib 100 mg once daily and continue on study treatment until evidence of disease progression, death, or unacceptable adverse events.
  Interventions: Drug: Buparlisib

INTERVENTIONS:
Drug: Buparlisib — Patients will receive oral buparlisib 100 mg once daily and continue on study treatment until evidence of disease progression, death, or unacceptable adverse events

SUMMARY:
The study will enrol adult female and male patients with BRAF wild-type melanoma and brain metastases who are not eligible for surgery or radiosurgery and failed prior therapy with ipilimumab, and patients with BRAF V600 mutation-positive melanoma and brain metastases who are not eligible for surgery or radiosurgery and who failed prior therapy with a BRAF inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
2. Patient has adequate bone marrow and organ function as defined by the following laboratory values; (Clinical labs - performed within 14 days prior to enrolment)

   Hematology
   1. Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
   2. Platelet count ≥ 100 x 109/L (For patients with haematologic malignancies involving the bone marrow, platelet count > 75 x 109/L)
   3. Haemoglobin ≥ 9.0 g/dL Coagulation
   4. INR ≤ 1.5

   Biochemistry e. Potassium and calcium (corrected for albumin), within normal limits for the institution, or ≤ Grade 1 if judged not clinically significant by the investigator f. Serum creatinine ≤ 1.5 x ULN and/or creatinine clearance > 50% LLN (Lower Limit of Normal) g. Total Serum bilirubin ≤ ULN (or <1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome, which is defined as presence of several episodes of unconjugated hyperbilirubinemia with normal results from CBC count (including normal reticulocyte count and blood smear), normal liver function test results, and absence of other contributing disease processes at the time of diagnosis h. AST (SGOT) and ALT (SGPT) below or equal upper limit of normal range or (≤ 3.0 x ULN if liver metastases are present) i. Fasting plasma glucose (FPG) ≤ 120mg/dL or ≤ 6.7 mmol/L j. HbA1c ≤ 8%
3. Patient is able to swallow and retain oral medication
4. Patient must be at least 18 years old
5. Patient must have an estimated life expectancy > 8 weeks in the opinion of the investigator
6. Patient must have ECOG performance status < 2

   Nature of illness and treatment history
7. Histologically confirmed diagnosis of melanoma
8. Patient must has shown evidence for PD in the brain by MRI without leptomeningeal disease
9. Contrast enhanced brain MRI and CT for chest / abdomen / pelvis or MRI for abdomen / pelvis must be performed within 28 days before first dose of study treatment
10. Patient is able to be assessed by periodic MRI and CT scan
11. Patients BRAF V600 wildtype:

    * must have objective evidence of progressive disease during or
    * following treatment with anti-CTLA-4 containing therapy for advanced melanoma
12. Patients BRAF V600 mutation positive:

    - must have objective evidence of progression of disease during or
    * following treatment with a BRAF inhibitor
    * not be eligible for surgery or radiosurgery
13. Time interval between last day of previous anti-tumour local or systemic treatment and first dose of buparlisib:

    * 14 days elapsed from last treatment with surgery or radiosurgery
    * 28 days elapsed from last treatment with whole brain radiation
    * 28 days have elapsed from last dose of approved or investigational chemo-, cytokine-, immune-, biological-, or vaccine-therapy
14. Participants must have recovered to a grade 0 or 1 from the toxic effects of prior therapy

Exclusion Criteria:

1. Patient has a known hypersensitivity to any of the excipients of buparlisib
2. Patient who has received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered to Grade 1 or better from related side effects of such therapy (except alopecia)
3. Patient has not recovered to Grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
4. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects
5. Patient is currently receiving increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent;

   1. The following uses of corticosteroids are permitted: single doses; e.g. with standard premedication for taxanes; topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
   2. Patient taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, rufinamide carbamazepine, oxcarbazepine, eslicarbazepine, felbamate, and topiramate (only when daily dose exceeds 200 mg). Participant must be off any EIAEDs for at least two weeks prior to starting study
   3. Requirement of more than 4 mg dexamethasone daily
6. Patient is being treated at start of study treatment with any of the following drugs:

   1. Drugs known to be strong inhibitors or inducers of isoenzyme CYP3A including herbal medications.
   2. Drugs with a known risk to induce Torsades de Pointes
   3. Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to starting study treatment is allowed.
   4. Patient who has received prior treatment with a PI3K inhibitor, AKT inhibitor or mTOR inhibitor
   5. Patient who have received anti-angiogenic or anti-VEGF targeted agents
7. Patient is currently receiving warfarin or any other coumarin-derivative anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
8. Patient who has who have other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study (e.g., active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
9. Patient has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory)
10. Patient has any of the following cardiac abnormalities:

    a. symptomatic congestive heart failure
    1. history of documents congestive heart failure (New York Heart Association NYHA functional classification III-IV, see Appendix 6), Documented cardiomyopathy
    2. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)

    b. Myocardial infarction < 6 months prior to enrolment c. unstable angina pectoris d. serious uncontrolled cardiac arrhythmia e. Symptomatic pericarditis f. QTcF > 450 msec on the screening ECG (using the QTcF formula) g. Currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
12. Participants with the following mood disorders as judged by the Investigator or a psychiatrist, or as result of participant's mood assessment questionnaire:

    a. Patient has a score of ≥ 12 in the PHQ-9 questionnaire, see Appendix 7 b. Patient selects a response of '1, 2, or 3' to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9) c. Patient has GAD mood scale score of ≥ 15 d. Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.

    e. Patient has anxiety ≥ CTCAE grade 3
13. Patient has other prior or concurrent malignancy (except for the following adequately treated basal cell or squamous cell skin cancer , or GI cancer resected completely by endoscopy procedures or any other cancer from which the patient has been disease free for ≥ 3 years)
14. Patient has a history of non-compliance to medical regimen or inability to grant consent
15. Patient is concurrently using other approved or investigational antineoplastic agent.
16. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL). Patients with elevated hCG at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5-7 days later, or pregnancy has been ruled out by vaginal ultrasound
17. Patient who does not apply highly effective contraception during during the study and through the duration as defined below after the final dose of study treatment:

    a. Sexually active males should use a condom during intercourse while taking drug and for 16 weeks after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

    b. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 4 weeks after the final dose of study treatment c. Highly effective contraception is defined as either: i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient] iv. Use a combination of the following (both a+b):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/ film/ cream/vaginal suppository.
3. Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as buparlisib decreases the effectiveness of hormonal contraceptives.

Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

For women with therapy-induced amenorrhea, oophorectomy or serial measurements of FSH and/or estradiol are needed to ensure postmenopausal status.

NOTE: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.

18. Patient with poorly controlled diabetes mellitus (glycosolated hemoglobin > 8%) or poorly controlled steroid-induced diabetes mellitus (glycosolated hemoglobin > 8%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Intracranial disease control rate | 6 weeks
  Intracranial disease control rate - defined as the percentage of patients whose intracranial response is a confirmed complete response, partial response or stable disease assessed by investigators using modified RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall response rate | 12 weeks
Duration of response for the subsets of patients with confirmed intracranial CR or PR | Up to 60 weeks
Duration of response for the subsets of patients with confirmed overall CR or PR | Up to 60 weeks
Progression free survival | week 24
Overall survival | week 52
Number of Adverse Events | Up to 104 weeks
  e.g. clinically significant laboratory abnormalities, vital signs, ECG, ECHO and clinical monitoring/observation.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Dermatology, University Hopsital, Dresden
  - Department of Dermatology, University Hospital, Tübingen